CLINICAL TRIAL: NCT00977704
Title: An Open-label Study of the Safety of Restylane and Perlane in the Correction of Peri-oral Wrinkles.
Brief Title: Study of Restylane and Perlane in the Correction of Peri-Oral Wrinkles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medicis Global Service Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-1900-01
Record Dates: First submitted 2009-09-14; First posted 2009-09-16 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-05

CONDITIONS: Peri-oral Wrinkles
Keywords: Correction of peri-oral wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Restylane and Perlane (Active Comparator): Restylane and Perlane administered by injection. Recommended volume of 6.0 mL. Injection on study day 1 with an optional touch up on study day 14.
  Interventions: Device: Restylane and Perlane

INTERVENTIONS:
Device: Restylane and Perlane

SUMMARY:
This is an open-label study to assess safety using Restylane and Perlane in the correction of facial wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Same Wrinkle Severity (either both Moderate [3] or both Severe [4]) of marionette lines and upper peri-oral rhytids

Exclusion Criteria:

* Active or chronic skin disease, inflammation or related conditions, near or on the Nasolabial Folds
* Subjects who had undergone procedures based on active dermal response (e.g., laser or chemical peeling procedures) within 6 months prior to study entry
* Use of any facial tissue augmenting therapy with non-permanent filler or aesthetic facial surgical therapy within 9 months prior to study entry
* Permanent implant placed in the Nasolabial Fold area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sanstead, RN, BSN, CCRC, Study Chair — Medicis Global Services
Locations (2):
- United States (2):
  - Call For Information, Coral Gables, Florida
  - Call For Information, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Perlane and Restylane: Perlane and Restylane used open label to correct peri-oral wrinkles
Period: Overall Study
Arm/Group | Perlane and Restylane
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Perlane and Restylane
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 59.6 (4.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Local and Systemic Adverse Events
Description: To examine the safety of Restylane and Perlane when used in the treatment of facial wrinkles and folds by identification of the point incidence of:
  * All local adverse events as reported by healthcare professional
  * All systemic adverse events (related and unrelated)
Time Frame: 2-weeks
Population: Primary object is to examine safety using descriptive statistics (frequency and percentage). Analysis was on the Intent to treat Population of all treated subjects, including those subjects for whom only incomplete data were available. No considerations (e.g. imputation) were made for missing data.
Measure: Number; unit: percentage of participants
Groups:
- Restylane and Perlane: Single arm safety study of subjects receiving Restylane and Perlane.
Arm/Group | Restylane and Perlane
Number analyzed (Participants) | 20
percentage of participants | 100

ADVERSE EVENTS:
Arm/Group | Perlane and Restylane
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perlane and Restylane (N=20)
Bruising (General disorders) | 19 (27)
Tenderness (General disorders) | 10 (20)
Swelling (General disorders) | 8 (11)
Redness (General disorders) | 4 (5)
Headache (Nervous system disorders) | 2 (2)
Discomfort (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Researcher agree to submit to Medicis for Medicis' prior review and written approval, which approval shall not be unreasonably withheld, any written publication utilizing results or other data generated from this study at least ninety days, or, for abstracts, at least thirty days before such publication is presented or submitted for publication.